CLINICAL TRIAL: NCT00092144
Title: A Multicenter, Double-Blind, Placebo-Controlled, Randomized, Parallel-Group Study to Evaluate the Clinical Effect of Oral MK0476 Vs Placebo During the Allergy Season in Patients With Seasonal Aeroallergen Sensitivity and Chronic Asthma Which is Also Active During Allergy Season
Brief Title: Study of an Approved Drug in Patients With Asthma (0476-289)(COMPLETED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0476-289; 2004_028
Record Dates: First submitted 2004-09-21; First posted 2004-09-24 (Estimated); Last update posted 2024-08-15 (Actual); Status verified 2022-01

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — montelukast; Duration of Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: MK0476, montelukast sodium / Duration of Treatment: 4 weeks
Drug: Comparator: placebo / Duration of Treatment: 4 weeks

SUMMARY:
The purpose of this study is to assess the efficacy and safety of an approved drug on asthma symptoms in patients with chronic asthma which is also active during the allergy season.

ELIGIBILITY:
Inclusion Criteria:

* Asthma symptoms brought on by allergies

Exclusion Criteria:

* Patient has any lung disease
* Currently have a sinus infection or cold symptoms

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2004-02-26 (Actual); Primary Completion 2004-06-15 (Actual); Study Completion 2004-06-15 (Actual)

PRIMARY OUTCOMES:
To assess daytime asthma symptoms as measured by daily diaries over a 3-week treatment period

SECONDARY OUTCOMES:
To assess the following over a 3-week treatment period:
nighttime symptoms
AM PEFR
PM PEFR
B-agonist use
asthma attacks
discontinuations due to asthma

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Busse WW, Casale TB, Dykewicz MS, Meltzer EO, Bird SR, Hustad CM, Grant E, Zeldin RK, Edelman JM. Efficacy of montelukast during the allergy season in patients with chronic asthma and seasonal aeroallergen sensitivity. Ann Allergy Asthma Immunol. 2006 Jan;96(1):60-8. doi: 10.1016/S1081-1206(10)61041-1. PMID 16440534